CLINICAL TRIAL: NCT03469193
Title: Evaluation Protocol of the Installation of Knee Unicompartmental Prosthesis (Journey (Smith & Nephew)) With Mechanical Ancillary Versus Robotic Assisted (Navio System). Prospective, Monocentric, Randomized, Open Label Study.
Brief Title: Evaluation Protocol of the Installation of Knee Unicompartmental Prosthesis (Journey (Smith & Nephew)) With Mechanical Ancillary Versus Robotic Assisted (Navio System).
Acronym: PUC NAVIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0512; 2017-A03292-51 (Other: ANSM)
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis Of Knee
Keywords: knee unicompartmental prosthesis; KneeKG system; robotic-assisted; alignment; implants positioning; International Knee Society; Forgotten joint score
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal PUC implanted with mechanical ancillary (Active Comparator)
  Interventions: Procedure: internal PUC implanted with mechanical ancillary
- Internal PUC implanted with robotic assistance (Experimental)
  Interventions: Procedure: Internal PUC implanted with robotic assistance

INTERVENTIONS:
Procedure: internal PUC implanted with mechanical ancillary — The control group consists of patients operated with a mechanical ancillary (reference surgery in our department). In this technique, bone sections are made with a standardized ancillary (manually adjusted bone cutting guides), according to preoperative radiological planning. The positioning of the implants is done manually and controlled by the placement of test implants.
  Arms: internal PUC implanted with mechanical ancillary
Procedure: Internal PUC implanted with robotic assistance — Patients are operated by robotics (surgery that we want to develop systematically in our service). 3D modeling of the knee allows the operator to perform a dynamic planning taking into account the reducibility of the deformation and the model of the implant. The operator can position the implants in three dimensions of the space without difficulty. This makes it possible to visualize, before the bone resections, the angular correction obtained between 0 and 130° flexion and alignment of the prosthesis by visualizing the contact points between the two implants. Bone resections will be performed using a guided retro bone drill. The system retracts more or less the cutter according to the bone thickness to be removed. This technique requires the insertion of two threaded plugs in the tibia and two in the femur to position the sensors that will allow the acquisition of anatomical landmarks of the lower limb and then 3D modeling
  Arms: Internal PUC implanted with robotic assistance

SUMMARY:
Unicompartmental knee arthroplasty by unicompartmental prosthesis (PUC) is a treatment for isolated internal femoro-tibial osteoarthritis. This intervention is justified in cases of significant discomfort, failure of medical treatment and the absence of osteoarthritis in femoro tibial external and patellofemoral femoro compartments. It aims to replace the native internal femoral tibial articulation by a joint between two implants, without intervening on the other compartments. The functional results of PUC are superior and faster than those obtained with total knee arthroplasty (TKA). Its indications and its realization are on the other hand very demanding to allow an optimal functional result.

Robotic-assisted surgery provides an excellent level of precision, which could allow better positioning of implants, compared to the use of a mechanical ancillary, according to the first published studies. The functional results and survival of these implants could also be improved.

The internal PUC with mechanical ancillary is carried out for many years in the orthopedic surgery department of Croix Rousse. For 3 years this surgery is sometimes performed with robotic assistance.

The investigators would like to prospectively evaluate the clinical and radiological impact of robotic-assisted surgery when performing a Journey unicompartmental prosthesis (Smith & Nephew).

The assessment of alignment during walking seems to be a paramount parameter in the results of the PUC and has not so far been evaluated in this type of robotic-assisted surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult (age ≥ 18 years)
* Diagnosis of unicompartmental knee osteoarthritis ( osteoarthritis internal femoral tibial (AFTI))
* Indication of unicompartmental knee arthroplasty of first intention posed

Exclusion Criteria:

* History of femoral or tibial osteotomy of valgization or varisation
* Reconstruction of the associated cruciate ligament
* Refusal to participate in the study
* Pregnant women, parturient or nursing mothers
* Persons deprived of their liberty by a judicial decision or administrative staff, persons under psychiatric care, persons admitted to a health or social institution to other purposes.
* Major persons subject to a legal protection measure or unable to express their consent
* Patient not affiliated to a social security scheme
* Patient participating in another interventional research excluding routine care research (former regulation) and category 2 searches not interfering with criterion analysis main

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
proportion of patients with Angle Hip Knee Ankle (HKA) (lower limb axis) restitution at 178 ° +/- 2 ° when the foot is touched with the floor and during the single support phase. | At 6 month postsurgery
  This criterion will be measured using a KneeKG system for dynamic analysis of knee movements.
  This system is non-invasive, non-radiating, non-painful. It is a dynamic tibiofemoral tracing device by infrared camera validated. The KneeKG system will be used according to its instructions for use.

SECONDARY OUTCOMES:
Radiological positioning of implants | At 6 month and 24 month postsurgery
  Measurements of HKA, frontal alignment of tibial and femoral implants, sagittal alignment of the femoral implant, tibial implant slope and the presence of peri-prosthetic edgings will be performed on a Standard radiography of the knee operated from the front, in profile and on a standing pangonometry
Comparison of the means of the International Knee Society (IKS) overall score between the groups. | At 6 month and 24 month postsurgery
  This is the international benchmark for clinical and functional evaluation in knee surgery. The 2011 version provides a more accurate, complete and comprehensive vision than the previous version.
Comparison of the Forgotten Joint Score | At 6 month and 24 month postsurgery
  The Forgotten score helps to analyze the patient's attention to the fact that his articulation has been replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Lustig, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Batailler C, Lording T, Naaim A, Servien E, Cheze L, Lustig S. No difference of gait parameters in patients with image-free robotic-assisted medial unicompartmental knee arthroplasty compared to a conventional technique: early results of a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):803-813. doi: 10.1007/s00167-021-06560-5. Epub 2021 Apr 11. PMID 33839803